CLINICAL TRIAL: NCT03366636
Title: Project Legacy Impact Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: ETR Associates (Other)
Responsible Party: Principal Investigator, Mona Desai, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHLA-17-00322
Record Dates: First submitted 2017-11-17; First posted 2017-12-08 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy Prevention; Sexual Behavior; Contraception Behavior; Sexually Transmitted Diseases
Keywords: Pregnancy Prevention; Adolescents; STIs/STDs; Self-sufficiency
MeSH Terms: conditions — Sexual Behavior; Contraception Behavior; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control/comparison group will be receiving only their usual services which are offered at the agencies they frequent, including mental health services, case management, job training, educational services, and, in specific venue contexts, may receive HIV risk reduction or other "sex education" interventions such as Street Smart. These same services are also open to the intervention group. Usage of these services varies by site (residential vs drop-in; city (San Diego vs Los Angeles) and type of service (case management, mental health, health care, etc.).
- Project Legacy (Experimental): The experimental/intervention arm will receive the Project Legacy intervention
  Interventions: Behavioral: Project Legacy

INTERVENTIONS:
Behavioral: Project Legacy — Project Legacy - Project Legacy is a 5-week, twice a week, 10 sessions small group intervention that encourages homeless and at-risk of homeless youth ages 14-19 to imagine a positive future and discuss how current risk behaviors can be a barrier to a successful adulthood. The program includes thinking about the future, the importance of positive social supports, short and long-term goal planning, and decision making. The program also includes life skills building, addressing past and current risk behaviors, linking to resources and navigating service systems, information on contraception and condoms, a healthy life plan and self-sufficiency. The 5 content core elements are the following:
  * 1. Thinking about the future
  * 2. Present actions to achieve future success
  * 3. Safeguarding one's future
  * 4. Creating a Healthy Life Plan
  * 5. Navigating service systems
  Arms: Project Legacy

SUMMARY:
This study will design and rigorously evaluate the efficacy of Project Legacy, a five week positive youth development intervention to decrease sexual risk for unintended pregnancies and STIs among youth experiencing homelessness or at risk of homelessness aged 14-19. This randomized control trial will compare Project Legacy to a usual services control.

DETAILED DESCRIPTION:
The study uses a multi-site randomized group trial (RGT) cohort design to evaluate the Project Legacy intervention curriculum for reducing sexual risk behaviors among homeless youth age 14-19. CHLA project staff will work with 6 homeless youth serving sites in Southern California (Los Angeles, San Diego) to recruit 600 youth. Randomization to the intervention or control condition will occur at the group level and will be stratified by site. Field staff will survey all eligible homeless youth who provide consent to participate in the study at baseline (before randomization and implementation) and at 3 and 9 months post intervention (5-5.5 and 11-11.5 months post-baseline). The program group will receive an additional intervention-based survey immediately upon completion of the program.

Youth in the control condition will receive the normal standard of care provided at the recruitment sites. Services available as standard of care at the recruitment sites include: medical care; mental health services; substance abuse services; educational, career, and vocational services. Intervention participants will not be excluded from receiving these services as well. Surveys will capture mental and physical health care service utilization and services to reduce substance use across both groups. The study team will monitor HIV and pregnancy prevention programming and other similar goal-planning/decision-making interventions offered to homeless youth in the study areas during the program implementation and follow-up period via interviews with site staff. The study team will include selected program exposure items on the follow up surveys to assess youth's self-reported exposure to similar goal-planning/decision-making and sexual health (pregnancy prevention and STI/HIV) education.

ELIGIBILITY:
Inclusion Criteria:

* Served or identified on outreach by one of our partner homeless youth serving agencies in Los Angeles or San Diego
* 14-19 years of age
* English-language speaker (able to complete consent and survey in English)
* not currently pregnant
* no immediate travel plans (are planning on being in the area for the length of the intervention - 8 weeks).

Exclusion Criteria:

* Outside of age range
* Currently pregnant
* Not planning to be in the area for the length of the intervention
* Previously enrolled in the study

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 571 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline lack of consistent current use (<80%) of contraception (including condoms) at 11 months | Assessed at baseline and 11 months post-baseline
  Current use of contraception (including condoms) is defined as using contraception at >80% of instances of vaginal intercourse in the past 3 months.
Change from baseline in current vaginal and anal sex without condom at 11 months | Assessed at baseline and 11 months post-baseline
  This outcome measure is defined as the proportion of instances of vaginal and anal sex without a condom in the past 3 months.

SECONDARY OUTCOMES:
Sexual initiation / activity (vaginal) | Assessed at baseline, 5 months post-baseline, and 11 months post-baseline
  Ever engaged in vaginal sex.
Current birth control use (vaginal sex) | Assessed at baseline, 5 months post-baseline, and 11 months post-baseline
  Current birth control use is defined as the number of instances of vaginal sex during which contraception was used (including condoms) in the past 3 months.
Current condom use (vaginal sex) | Assessed at baseline, 5 months post-baseline, and 11 months post-baseline
  Current condom use for vaginal sex is defined as: the number of instances of vaginal sex during which condoms were used in the past 3 months
Proportion of youth who have vaginal intercourse without the consistent use of contraception | Assessed at baseline, 5 months post-baseline, and 11 months post-baseline
  This outcome is defined as using contraception for less than 80% of instances of vaginal sex in the past 3 months.
  1. "In the past 3 months, how many times did you have vaginal sex?"
  2. "When you had vaginal sex in the past 3 months, how many times did you and your partner(s) have sex and NOT use any type of contraception (in other words, EITHER a condom OR other method of birth control)? By birth control, we mean using condom, birth control pills, the shot, the patch, the ring, IUD, or implant".
Current contraception use (among females) | Assessed at baseline, 5 months post-baseline, and 11 months post-baseline
  Current contraception use is defined as the use of one or more methods of effective contraception in the past 3 months
Current marijuana or alcohol use | Assessed at baseline, 5 months post-baseline, and 11 months post-baseline
  Current marijuana or alcohol use is defined as marijuana or alcohol use in the past 3 months
Stable living environment at the time of the follow-up (current) | Assessed at baseline, 5 months post-baseline, and 11 months post-baseline
  Stable living defined as living in a parents', relatives' or foster parents' home; a group home or residential facility or a tenant of an apartment.
Employment experience (current) | Assessed at baseline, 5 months post-baseline, and 11 months post-baseline
  Employed part or full-time since baseline; certificate, post-high school or college completed;
Engagement in job-readiness services | Assessed at baseline, 5 months post-baseline, and 11 months post-baseline
  Services defined as job preparedness skill-building, job internships, or educational services
Social support (current) | Assessed at baseline, 5 months post-baseline, and 11 months post-baseline
  Social support is measured using The Multidimensional Scale of Perceived Social Support. Total scores range from 7 to 84 and each subscale score ranges from 4 to 28, with a higher score indicating greater social support. which are averaged together to get the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie F Clark, PhD, MPH, Principal Investigator — University of Southern California
Locations (12):
- United States (12):
  - Five Keys, Boyle Heights, California
  - Youth Program, Long Beach, California
  - Century Villages at Cabrillo, Long Beach, California
  - Da Vinci Rise High, Los Angeles, California
  - LA CAUSA Youth Build, Los Angeles, California
  - Covenant House, Los Angeles, California
  - Los Angeles LGBT Center, Los Angeles, California
  - YMCA of San Diego County, Oceanside, California
  - San Diego Central Library, San Diego, California
  - San Diego Youth Services, San Diego, California
  - Monarch School, San Diego, California
  - Safe Place for Youth, Venice, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Rosa CJ, Montgomery SB, Kipke MD, Iverson E, Ma JL, Unger JB. Service utilization among homeless and runaway youth in Los Angeles, California: rates and reasons. J Adolesc Health. 1999 Mar;24(3):190-200. doi: 10.1016/s1054-139x(98)00081-0. PMID 10195802
- [Background] Edidin JP, Ganim Z, Hunter SJ, Karnik NS. The mental and physical health of homeless youth: a literature review. Child Psychiatry Hum Dev. 2012 Jun;43(3):354-75. doi: 10.1007/s10578-011-0270-1. PMID 22120422
- [Background] Rotheram-Borus MJ, Song J, Gwadz M, Lee M, Van Rossem R, Koopman C. Reductions in HIV risk among runaway youth. Prev Sci. 2003 Sep;4(3):173-87. doi: 10.1023/a:1024697706033. PMID 12940468
- [Background] Tucker JS, Sussell J, Golinelli D, Zhou A, Kennedy DP, Wenzel SL. Understanding pregnancy-related attitudes and behaviors: a mixed-methods study of homeless youth. Perspect Sex Reprod Health. 2012 Dec;44(4):252-61. doi: 10.1363/4425212. Epub 2012 Nov 13. PMID 23231333
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Chen P, Vazsonyi AT. Future orientation, impulsivity, and problem behaviors: a longitudinal moderation model. Dev Psychol. 2011 Nov;47(6):1633-45. doi: 10.1037/a0025327. Epub 2011 Sep 5. PMID 21895358
- [Background] Oyserman D, Terry K, Bybee D. A possible selves intervention to enhance school involvement. J Adolesc. 2002 Jun;25(3):313-26. doi: 10.1006/jado.2002.0474. PMID 12128042
- [Background] Thompson, S., Pollio, D., Constantine, J., Reid, D., Nebbitt, V. Short-term outcomes of youth receiving runaway and homeless shelter services. Research on Social Work Practice. 2002 Sept; 12: 589-603
- [Background] Juntunen, C.L., & Wettersten, K. Work hope: Development and initial validation of a measure. Journal of Counseling Psychology. 2006; 53(1): 94-106.
- [Background] Robitschek, C. Personal growth initiative: The construct and its measure. Measurement & Evaluation in Counseling & Development: American Counseling Association. 1998; 30(4): 183-198.
- [Background] Strauman, T.J. (2006). Adolescent Regulatory Focus Questionnaire. Unpublished questionnaire, Duke University, Durham, NC.
- [Background] Rice E, Milburn NG, Monro W. Social networking technology, social network composition, and reductions in substance use among homeless adolescents. Prev Sci. 2011 Mar;12(1):80-8. doi: 10.1007/s11121-010-0191-4. PMID 21194011
- [Background] Hansen WB, Paskett ED, Carter LJ. The Adolescent Sexual Activity Index (ASAI): a standardized strategy for measuring interpersonal heterosexual behaviors among youth. Health Educ Res. 1999 Aug;14(4):485-90. doi: 10.1093/her/14.4.485. PMID 10557519
- [Background] Trussell J. Contraceptive failure in the United States. Contraception. 2011 May;83(5):397-404. doi: 10.1016/j.contraception.2011.01.021. Epub 2011 Mar 12. PMID 21477680
- [Background] Oyserman D, Bybee D, Terry K, & Hart-Johnson T. Possible selves as roadmaps. Journal of Research in Personality 38: 130-149, 2004.
- [Background] Higgins ET. Beyond pleasure and pain. Am Psychol. 1997 Dec;52(12):1280-300. doi: 10.1037//0003-066x.52.12.1280. PMID 9414606